CLINICAL TRIAL: NCT04468503
Title: Comparative Effect of Protein Prescription Strategies on Nitrogen Balance and Upshots in Critically Ill Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Allama Iqbal Open University Islamabad (Other)
Collaborators: Shifa International Hospital (Other)
Responsible Party: Principal Investigator, Zainab Bibi, Prinicipal Investigator, Allama Iqbal Open University Islamabad
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: HEC acadmic research
Record Dates: First submitted 2020-07-03; First posted 2020-07-13 (Actual); Last update posted 2024-06-11 (Actual); Status verified 2024-06

CONDITIONS: Critical Illness; Malnutrition; Protein
Keywords: critical illness; protein; malnutrition
MeSH Terms: conditions — Critical Illness; Malnutrition

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 1 g per kg body weight per day (Active Comparator): Protein will be receive by patients that is 1g per kg per day, Patients will be assess and according to patient actual dry weight 1 g per kg of that weight protein will provided, energy will be provided according to ASPEN guideline 2016.
  Base line characters(BMI, nitrogen Balance, Protein biomarker, LFTs, RFTs, GCS)
  Interventions: Other: Two differnt protien prescription (ig per kg per day and 2g per kg /day )will be assigned to each group interventional
- 2 g per kg body weight per day (Active Comparator): Protein will be receive by patients that is 2g per kg per day, Patients will be assess and according to patient actual dry weight 1 g per kg of that weight protein will provided, energy will be provided according to ASPEN guideline 2016.
  Base line characters(BMI, nitrogen Balance, Protein bio marker, LFTs. , RFTs, GCS)
  Interventions: Other: Two differnt protien prescription (ig per kg per day and 2g per kg /day )will be assigned to each group interventional

INTERVENTIONS:
Other: Two differnt protien prescription (ig per kg per day and 2g per kg /day )will be assigned to each group interventional — In this study intervention will be the dose of protein, one group will be prescribed with the protein dose (1 g/kg/day) and other group will be on prescribed higher dose (2gm/kg/day) of protein according to the ASPEN guideline for critically ill and the energy requirements (other than proteins) will be 25 kcal/kg of adjusted body weight (Picolo et al.,). Each subject in the trail will provide remaining medical nutrition therapy according to the therapeutic guidelines in the field. The medical nutrition management other than protein will be adjust according to need of each patient.

SUMMARY:
This is Interventional clinical trail will be conducted in Internationale hospital ICU s patients with higher nutrition risk. two doses of protein 1 g/kg/day Vs 2 g/ kg day will be given and its outcome will be checked on nitrogen balance , clinical outcome length of hospital stay, mortality ratio and re admission within 30 days.

DETAILED DESCRIPTION:
STUDY DESIGN This is the prospective interventional randomized controlled trial in which effect of protein prescription on UUN and clinical outcome of critically ill patients enroll in the study will compare The NUTRIC scores will be calculated manually, based on data from the medical records of critically ill patients.This trail will be conducted in three stages.

In Phase I all admitted patients in critical care unit will be screen by. APACHE II NUTRIC Score Phase II: Patients with nutrition risk will randomly divided into two group (1:1) Interventional Group None Interventional Group Phase III: Follow the patient for 28 days after discharge from Hospital. Study Locale The study will be conducted in the ICUs (SICUs, MICUs, HDU) of Hospital in Islamabad, for this study organizational approval from formal ethical committee will be taken during the time period of six months.

STATISTICAL METHODS:

Descriptive statistics will be use for demographic data and over all outcomes, further more analytical stat will be used to the type of variables and objective of the study. Z test will be use for the comparison of quantitative variables and Chi square test will be use for categorical data. A NOVA will be use where applicable

.

ELIGIBILITY:
Inclusion Criteria:

Critically ill patient with nutritional risk Age >18 years Pt. ICU stay> 48hours

Exclusion Criteria:

Patients on ventilator > 72 hours < 48 hours.' stay in ICU Withdrawal of life support within 7 days of randomization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Urine Urea Nitrogen (UUN) for Nitrogen Balanace (NB) | for base line is within 24hours of randomization,for nitrogen balence reassessment every 72 hourly
  change in nitrogen balance from baseline.
Readmission in hospital within 30 days of discharge. | 30 days after discharge
  Patient will be followed for 30 days after discharge from hospital for monitoring, e.g. readmission in hospital Mortality ratio

SECONDARY OUTCOMES:
Sequential Organ Failure Assessment (SOFA Score) | up to 72 hours in ICU stay
  this tool will be use to track a person's status during the stay in an critical care unit (ICU) to determine the extent of a person's organ function or rate of failure, with a minimum SOFA score of 0 (most survival) and a maximum SOFA score of 24(risk of survival).
protein bio markers | up to 72 hours in ICU stay
  Blood Urea Nitrogen, Albumin, C- reactive protien

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Mahpara Safdar, phd, Study Chair — Allama Iqbal Open University
Locations (1):
- Allama Iqbal Open University, Islamabad, Federal, Pakistan

IPD SHARING:
Plan to Share IPD: No
basic detail

REFERENCES:
- [Derived] Bibi Z, Safdar M, Hadayat A. Comparative effect of protein dosage on nitrogen balance and health outcomes in critically ill patients. J Pak Med Assoc. 2025 May;75(5):699-703. doi: 10.47391/JPMA.20753. PMID 40500809